CLINICAL TRIAL: NCT01987544
Title: German: Effekte Eines Telemonitorisch überwachten Ergometertrainings Bei Patienten Mit Einer COPD Nach Exazerbation: Eine Prospektiv Randomisierte Studie
Brief Title: Effects of Ergometer Training With Telemonitoring in Patients With Chronic Obstructive Pulmonary Disease (COPD) After Exacerbation
Acronym: COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut für Pneumologie Hagen Ambrock eV (Industry)
Collaborators: Vitaphone GmbH (Unknown)
Responsible Party: Principal Investigator, Karl Josef Franke, Senior Physician Helios Klinik Hagen, Klinik für Pneumologie, Institut für Pneumologie Hagen Ambrock eV
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Telebike2013
Record Dates: First submitted 2013-11-13; First posted 2013-11-19 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2016-02

CONDITIONS: COPD
Keywords: COPD; telemonitoring; training; ergometer; telemedicine
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Information Motivation Behavioral Skills Model

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Self-Control (Active Comparator): 3 months of ergometer training under self control at home without any interventional motivation.
  Interventions: Other: Ergometer Training
- Motivation (Experimental): 3 months of ergometer training at home with telemonitoring and motivation phone calls once a week when training sessions drop below 20 minutes per day.
  Interventions: Other: Ergometer Training; Other: Motivation

INTERVENTIONS:
Other: Ergometer Training
  Other Names: Ergometer
Other: Motivation
  Other Names: Telemonitoring; Phone Calls
  Arms: Motivation

SUMMARY:
Home ergometer training combined with online monitoring and regular telephone support could prove to be a cost-effective method to improve physical performance and quality of life in COPD patients.

The primary objective of the study is to demonstrate a significantly higher daily workout time in patients that are monitored during home ergometer training with telephone support compared to conventional home ergometer training. Consequently we expect an increased quality of life related to the illness and a decreasing BODE-Index. A post-interventional lower BODE-Index correlates with a reduced risk of hospitalisation and mortality.

DETAILED DESCRIPTION:
Hypothesis: There will be an increased prevalence, morbidity and mortality of COPD during the next decades. On the other hand there is a clear correlation between life expectancy and physical activity in this disease. Telemedicine concepts promise new treatment strategies with favourable impact on the long-term process of COPD.

ELIGIBILITY:
Inclusion Criteria:

* COPD

Exclusion Criteria:

* tumor diseases
* unstable coronary heart disease
* untreated cardiac valve disease
* incapable of giving consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2012-09; Primary Completion 2014-12 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Training time | 3 month
  Patients workout at home with a provided bicycle ergometer, the daily training target is 30 minutes. The training time is monitored online using a GSM module.

SECONDARY OUTCOMES:
BODE-Index | 3 month
  The BODE-Index is a grading tool to assess the progress of COPD with a range of 0 to 10 points. A post-interventional lower BODE-Index correlates with a reduced risk of hospitalisation and mortality.

OTHER OUTCOMES:
CAT (COPD Assessment Test) | 3 month
  The CAT is a questionnaire to measure the impact of COPD on a person's life. The range is 0 to 40 points.

CONTACTS AND LOCATIONS:
Locations (1):
- Helios Klinik Hagen, Hagen, North Rhine-Westphalia, Germany

REFERENCES:
- [Derived] Cox NS, Dal Corso S, Hansen H, McDonald CF, Hill CJ, Zanaboni P, Alison JA, O'Halloran P, Macdonald H, Holland AE. Telerehabilitation for chronic respiratory disease. Cochrane Database Syst Rev. 2021 Jan 29;1(1):CD013040. doi: 10.1002/14651858.CD013040.pub2. PMID 33511633